CLINICAL TRIAL: NCT05143736
Title: Nasal and Gut Microbiota Combined Clinical Events Predicts the Prognosis of Patients With Sepsis: a Prospective, Multicentered, Diagnostic Trial
Brief Title: Nasal and Gut Microbiota Combined Clinical Events Predicts the Prognosis of Septic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Liu Zhanguo, Vice Director of Critical Care Medicine, Principal Investigator, Zhujiang Hospital
Other Study IDs: 2021-KY-108-01
Record Dates: First submitted 2021-10-16; First posted 2021-12-03 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-01

CONDITIONS: Sepsis; Septic Shock
Keywords: Sepsis; Septic Shock; nasal microbiota; gut microbiota
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Total DNA of nasal and gut microbiota coming from patients with sepsis will be extracted , amplified, and sequenced.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Modeling cohort: The population enrolled at the intensive care unit of Zhujiang Hospital of Southern Medical University in Guangdong Province, China will be used as a modeling cohort.For the patients in this cohort, the nasal and fecal specimens and related clinical information will collected to construct the prediction model.
  Interventions: Diagnostic Test: gut and nasal microbiota detection
- validation cohort: The population enrolled at the intensive care unit of Dongguan People's Hospital in Guangdong Province, China will be used as a validation cohort.
  Interventions: Diagnostic Test: gut and nasal microbiota detection

INTERVENTIONS:
Diagnostic Test: gut and nasal microbiota detection — The nasal and fecal specimens will be collected by swabs from subjects with sepsis. After that, total DNA of nasal and gut microbiota will be extracted , amplified, and sequenced to determine the gut and nasal microbiota.

SUMMARY:
In this prospective, multicentered , diagnostic trial, nasal and fecal specimens will collected from patients with sepsis in two critical care units(ICU) at the enrollment day ,the third, seventh, and fourteen days after enrollment or until ICU discharge (whatever come first). Total DNA from the nasal and fecal specimens will be extracted, amplified, and sequenced to determined the characteristics of gut microbiota and nasal microbiota. Finally, the characteristics of gut microbiota and nasal microbiota combined clinical information will be used to construct a prediction model to predict the prognosis of sepsis.

DETAILED DESCRIPTION:
Background:

Sepsis should be defined as life-threatening organ dysfunction caused by a dysregulated host response to infection, with high morbidity and mortality, and its total mortality is 10% to 52%. In sepsis, it is not clear sufficiently about the relationship between intestinal and nasal microbiota character and the development of the sepsis.The study aim to construct a prediction model to predict the prognosis and development of sepsis.

Purpose:

1. To construct a prediction model using nasal and gut microbiota combined with clinical events to predict the prognosis of patients with sepsis and development of sepsis.
2. Analyze the characteristics of nasal and gut microbiota in patients with sepsis using microbiology.

Methods:

nasal and fecal specimens will collected from patients with sepsis in two critical care units(ICU) at the enrollment day ,the third, seventh, and fourteen days after enrollment or until ICU discharge (whatever come first). Total DNA from the nasal and fecal specimens will be extracted, amplified, and sequenced to determined the characteristics of gut microbiota and nasal microbiota. Meanwhile, some related clinical information also will be collected,including demographic characteristics, comorbidities, infection site, results of the microbiology experiments, vital signs, invasive tubing indwelling at enrollment，combined medication，the requirement of organ function support, laboratory indexing, sequential organ failure assessment score and Acute Physiology and Chronic Health Evaluation score. Finally, the characteristics of gut microbiota and nasal microbiota combined the clinical information will be used to construct a prediction model to predict the prognosis of sepsis. The primary outcome is the 28-day all-cause mortality. The secondary outcomes are the incidence of septic shock, the incidence of persistent inflammation- immunosuppression catabolism syndrome and the 90-day all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the 2016 International Sepsis Guidelines diagnostic criteria (sepsis 3.0).
2. Serum procalcitonin≥ 2 ng/mL at enrollment.

Exclusion Criteria:

Patients will be excluded if participants meet any of the following criteria:

1. age<18 years old or > 80 years
2. pregnancy or lactation
3. solid organ or bone marrow transplant
4. advanced pulmonary fibrosis
5. HIV-positive
6. neutropenia;
7. hematological/lymphatic tumors have no remission;
8. limited care (lack of commitment to full and aggressive support);
9. long-term use of immunosuppressive drugs or immunodeficiency;
10. advanced tumors;
11. combined with noninfectious factors leading to death (uncontrolled large bleeding, cerebral hernia, etc.);
12. Combined with autoimmune diseases
13. Paraquat poisoning
14. Combined with Nasopharyngeal carcinoma
15. Combined with chronic nasosinusitis
16. Combined with severe nasal injuries

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In this study, patients who met the Sepsis 3.0 diagnostic criteria and with PCT ≥ 2ng/ml and will be recruited.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
All-cause death at 28 days | The outcome will be assessed on the 28th day from enrollment
  All-cause mortality from the enrollment to the 28th day

SECONDARY OUTCOMES:
Incidence of septic shock | The outcome will be assessed diurnally until ICU discharge，the longest evaluation duration is no more than 28 days
  Incidence of septic shock during the ICU stay.
Incidence of persistent inflammation-immunosuppression catabolism syndrome (PICS) | The outcome will be assessed diurnally until ICU discharge，the longest evaluation duration is no more than 28 days
  The incidence of PICS during the ICU stay. Patients who meet all the following diagnostic criteria will be diagnosed PICS: 1) the duration of ICU stay more than 14 days, 2) the level of serum C reactive protein > 50ug/dL, 3) Lymphocyte counts<0.80*10^9/L,4) serum albumin<3g/dL, 5) serum prealbumin<10mg/dL, 6) The creatinine height index<80%. 7)weight loss more than 18% or BMI<18

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Liu, M.D.PhD, Principal Investigator — Department of Critical Care Medicine of Zhujiang Hospital
Locations (2):
- China (2):
  - Department of Critical Care Medicine of Dongguan People's Hospital, Dongguan, Dongguan, Guangdong
  - Department of Critical Care Medicine of Zhujiang Hospital, Guanzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated and analyzed during the study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Tan XL, Liu HY, Long J, Jiang Z, Luo Y, Zhao X, Cai S, Zhong X, Cen Z, Su J, Zhou H. Septic patients in the intensive care unit present different nasal microbiotas. Future Microbiol. 2019 Mar;14(5):383-395. doi: 10.2217/fmb-2018-0349. Epub 2019 Feb 26. PMID 30803270